CLINICAL TRIAL: NCT00002912
Title: A PHASE I COOPERATIVE AGREEMENT PEDIATRIC TRIAL OF MITOXANTRONE, ETOPOSIDE AND PSC-833 (PSC-ME) THERAPY IN PATIENTS WITH RELAPSED AND REFRACTORY ACUTE LEUKEMIA
Brief Title: Combination Chemotherapy Plus PSC-833 in Treating Children With Refractory or Relapsed Acute Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01835; POG-9423; CCG-P9423; CDR0000065285 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 1999-11-01; First posted 2004-04-29 (Estimated); Last update posted 2013-02-01 (Estimated); Status verified 2010-08

CONDITIONS: Leukemia
Keywords: recurrent childhood acute lymphoblastic leukemia; recurrent childhood acute myeloid leukemia; secondary acute myeloid leukemia
MeSH Terms: conditions — Leukemia; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Etoposide; Mitoxantrone; valspodar

ARMS (1):
- Arm I (Experimental): Patients undergo induction therapy consisting of etoposide IV and mitoxantrone IV on days 1-5. Patients then receive PSC-833 IV over 124 hours beginning on day 2. A second course is administered no sooner than 21 days from the start of the first course if the marrow is hypocellular after the first course. Patients with persistent disease after 2 induction courses are removed from the study. Patients receive a total of 3 courses of etoposide/mitoxantrone. Patients who achieve complete remission after 1 induction course receive 2 courses of etoposide/mitoxantrone with PSC-833 as consolidation, beginning within 4 weeks of attainment of complete remission. Patients who achieve complete remission after 2 induction courses receive 1 course of etoposide/mitoxantrone with PSC-833 as consolidation. Cohorts of 3-6 patients receive escalating doses of PSC-833 until the maximum tolerated dose is determined. Patients are followed every 6 months.
  Interventions: Drug: etoposide; Drug: mitoxantrone hydrochloride; Drug: valspodar

INTERVENTIONS:
Drug: etoposide
Drug: mitoxantrone hydrochloride
Drug: valspodar

SUMMARY:
Phase I trial to study the effectiveness of PSC-833 plus etoposide and mitoxantrone in treating children who have refractory or relapsed acute leukemia. Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Some cancers become resistant to chemotherapy drugs. Combining PSC-833 with chemotherapy may reduce resistance to the drug and allow more cancer cells to be killed.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the maximum tolerated dose of PSC-833 in combination with mitoxantrone and etoposide in children with refractory or relapsed acute leukemia.

II. Determine the effects of PSC-833 on mitoxantrone and etoposide pharmacokinetics.

III. Quantify MDR1 gene expression and MDR1 P-glycoprotein expression and function in patient-derived leukemia cells.

OUTLINE: This is a dose escalation study of PSC-833.

Patients undergo induction therapy consisting of etoposide IV and mitoxantrone IV on days 1-5. Patients then receive PSC-833 IV over 124 hours beginning on day 2. A second course is administered no sooner than 21 days from the start of the first course if the marrow is hypocellular after the first course. Patients with persistent disease after 2 induction courses are removed from the study. Patients receive a total of 3 courses of etoposide/mitoxantrone. Patients who achieve complete remission after 1 induction course receive 2 courses of etoposide/mitoxantrone with PSC-833 as consolidation, beginning within 4 weeks of attainment of complete remission. Patients who achieve complete remission after 2 induction courses receive 1 course of etoposide/mitoxantrone with PSC-833 as consolidation. Cohorts of 3-6 patients receive escalating doses of PSC-833 until the maximum tolerated dose is determined. Patients are followed every 6 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Acute myeloid leukemia (AML) in one of the following categories:
* First relapse if initial CR less than 6 months
* Refractory to first or second induction with daunomycin, cytarabine, and thioguanine (DAT) or other anthracycline-containing regimens
* Relapse following bone marrow transplantation provided good trilineage engraftment followed transplant and greater than 6 months since transplant
* Presentation with secondary AML or AML evolving from myelodysplastic syndrome --Acute lymphocytic leukemia in one of the following categories:
* In second or subsequent relapse or failed second or later induction attempts regardless of prior remissions
* Relapsed following bone marrow transplantation provided good trilineage engraftment followed transplant and greater than 6 months since transplant
* No isolated CNS or extramedullary relapse

PATIENT CHARACTERISTICS:

* Age: Under 22 at diagnosis
* Performance status: Karnofsky 50-100% (ECOG 0-2)
* Lansky 40-100% (in patients under 12 years of age)
* Life expectancy: At least 8 weeks
* Bilirubin less than 1.5 mg/dL
* ALT less than twice normal
* Creatinine normal for age (within 2 standard deviations) OR glomular filtration rate at least 70 mL/min
* Albumin at least 3 g/dL
* Ejection fraction greater than 50% at rest or with 5% increase with exercise OR shortening fraction greater than 27% by echocardiogram
* No history of clinical heart failure
* No uncontrolled infection
* No anticonvulsant therapy
* No history of allergic reactions or anaphylaxis to etoposide not remediable by premedication
* Not pregnant or nursing
* Fertile patients must use effective contraception
* Third percentile weight for height

PRIOR CONCURRENT THERAPY:

* At least 4 weeks since chemotherapy and recovered
* Prior cumulative anthracycline dose no greater than 360 mg per square meter
* Hydroxyurea therapy allowed just prior to study for rapidly rising blast count

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 3 (Actual)
Dates: Start 1997-01; Primary Completion 2006-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary V.H. Dahl, MD, Study Chair — Lucile Packard Children's Hospital at Stanford University Medical Center
Locations (55):
- United States (50):
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - University of California San Diego Cancer Center, La Jolla, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - City of Hope National Medical Center, Los Angeles, California
  - Children's Hospital of Orange County, Orange, California
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - Stanford University Medical Center, Stanford, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - University of Florida Health Science Center, Gainesville, Florida
  - Emory University Hospital - Atlanta, Atlanta, Georgia
  - Robert H. Lurie Comprehensive Cancer Center, Northwestern University, Chicago, Illinois
  - Children's Memorial Hospital, Chicago, Chicago, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - University of Kansas Medical Center, Kansas City, Kansas
  - Johns Hopkins Oncology Center, Baltimore, Maryland
  - Boston Floating Hospital Infants and Children, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Children's Hospital of Michigan, Detroit, Michigan
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Children's Mercy Hospital, Kansas City, Missouri
  - Cardinal Glennon Children's Hospital, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - NYU School of Medicine's Kaplan Comprehensive Cancer Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Columbia Presbyterian Hospital, New York, New York
  - State University of New York - Upstate Medical University, Syracuse, New York
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Children's Hospital Medical Center - Cincinnati, Cincinnati, Ohio
  - Children's Hospital of Columbus, Columbus, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt Cancer Center, Nashville, Tennessee
  - Simmons Cancer Center - Dallas, Dallas, Texas
  - Cook Children's Medical Center - Fort Worth, Fort Worth, Texas
  - Texas Children's Cancer Center, Houston, Texas
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Primary Children's Medical Center, Salt Lake City, Utah
  - Children's Hospital and Regional Medical Center - Seattle, Seattle, Washington
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
  - Midwest Children's Cancer Center, Milwaukee, Wisconsin
- Australia (2):
  - Royal Children's Hospital, Parkville, Victoria
  - Princess Margaret Hospital for Children, Perth, Western Australia
- Canada (3):
  - Hospital for Sick Children, Toronto, Ontario
  - Montreal Children's Hospital, Montreal, Quebec
  - Hopital Sainte Justine, Montreal, Quebec

REFERENCES:
- [Result] O'Brien MM, Lacayo NJ, Lum BL, Kshirsagar S, Buck S, Ravindranath Y, Bernstein M, Weinstein H, Chang MN, Arceci RJ, Sikic BI, Dahl GV. Phase I study of valspodar (PSC-833) with mitoxantrone and etoposide in refractory and relapsed pediatric acute leukemia: a report from the Children's Oncology Group. Pediatr Blood Cancer. 2010 May;54(5):694-702. doi: 10.1002/pbc.22366. PMID 20209646
- [Result] Lacayo NJ, Lum BL, Chin DL, et al.: Pharmacokinetics of mitoxantrone in a Phase I Trial of PSC-833 (Valspodar) as an MDR1/Pg-P modulator in acute myeloid leukemia (AML) from the children's oncology group (COG). [Abstract] Proceedings of the American Society of Clinical Oncology 21: A-1583, 2002.